CLINICAL TRIAL: NCT04861337
Title: Effect of Remimazolam on Incidence of Postoperative Nausea and Vomiting Following General Anesthesia in High-risk Patients: a Multicenter, Double-blinded, Placebo-controlled Randomized Trial
Brief Title: Remimazolam and Postoperative Nausea and Vomiting in High-risk Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020-429
Record Dates: First submitted 2021-04-24; First posted 2021-04-27 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Postoperative Nausea and Vomiting; Benzodiazepine; High-risk Patients
Keywords: Postoperative nausea and vomiting; Benzodiazepines; High-risk patients
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — remimazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam Group (Experimental): Remimazolam infusion is initiated after induction of general anesthesia at a rate of 0.25 mg/kg/h and stopped 15 minutes before the end of surgery.
  Interventions: Drug: Remimazolam
- Placebo Group (Placebo Comparator): Placebo (0.9% saline) infusion is initiated after induction of general anesthesia at the same rate as in the remimazolam group and stopped 15 minutes before the end of surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Remimazolam — Remimazolam is infused at a rate of 0.25 mg/kg/h from end of anesthesia induction until 15 minutes before the end of surgery.
  Other Names: Remimazolam group
  Arms: Remimazolam Group
Drug: Placebo — Normal saline is infused at a rate same as in the remimazolam group from end of anesthesia induction until 15 minutes before the end of surgery.
  Other Names: Placebo group
  Arms: Placebo Group

SUMMARY:
This trial aims to explore whether the intraoperative use of remimazolam can reduce the incidence of postoperative nausea and vomiting (PONV) in high-risk patients. According to the Apfel's simplified score, patients with 3 or more of the following factors are at high risk of postoperative nausea and vomiting (PONV), i.e., women, non-smokers, history of PONV, and postoperative use of opioids.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is a common adverse event after general anesthesia. The incidence of PONV within 2 hours after surgery was approximately 14% in patients undergoing laparoscopic gynecological procedure and it could be about 22%-33% within 24 hours and as high as 80% in high-risk patients. Even with prophylaxis and treatment, such as 5-hydroxytryptamine 3 (5-HT3) receptor antagonists, the incidence of PONV is still about 7%-10%.

PONV is an important clinical problem that impact the recovery of patients. Firstly, it can be a highly distress experience to patients and reduce their satisfaction with medical services. Secondly, PONV is associated with prolonged stay in the postanesthesia care unit and hospital, and increase medical expenditures. Thirdly, PONV increases the risk of reflux aspiration and lung infection.

Risk factors for PONV in adults include anxiety, opioid use, and inflammation. A cohort study showed that patients with anxiety before surgery have a 5-fold increase in the risk of PONV. Opioids are one of the main causes of PONV, and the incidence of PONV increases with the increasing dose of opioids. Inflammation is also considered to be a potential molecular mechanism leading to PONV. Animal studies have shown that surgery can cause inflammation throughout the body and central nervous system, and stimulate the "vomiting center" , which leads to PONV.

Several clinical studies reported that midazolam decreased PONV. In a meta-analysis included 12 randomized trials (841 patients), the use of midazolam during the perioperative period reduced the risk of PONV by about 55%. Another Meta-analysis involving 16 randomized controlled studies also reported similar results. The use of midazolam during the perioperative period reduced the risk of PONV by approximately 45%.

The mechanism by which benzodiazepines reduce PONV is not fully understood, but may include the following. Benzodiazepines can reduce the incidence of anxiety and reduce the severity of anxiety. On the other hand, studies have shown that the use of remimazolam enhances the analgesic effect of remifentanil and may reduce the dose of opioids. Another aspect is benzodiazepines may suppress the inflammatory response.

Remimazolam is an ultra-short-acting benzodiazepine sedative. It has a more predictable fast onset, short duration of sedative action, and rapid recovery profile, but there is no clinical study on whether remimazolam has an effect on the incidence of PONV. The investigators speculate that remimazolam as a supplement anesthetic during general anesthesia can reduce the incidence of PONV.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Scheduled to undergo elective surgery under general anesthesia;
3. Judged to be at high risk of postoperative nausea and vomiting. According to the Apfel's simplified score, patients with 3 or more of the following factors are at high-risk: women, non-smokers, history of PONV, postoperative use of opioids.

Exclusion Criteria:

1. Refuse to participate;
2. Previous history of schizophrenia, epilepsy, Parkinson's disease or myasthenia gravis;
3. Severe liver dysfunction (Child-Pugh class C);
4. Severe renal dysfunction (dialysis required);
5. Patients of the American Society of Anesthesiologists (ASA) grade 4 and above;
6. Emergency surgery;
7. Continuously taking benzodiazepines for more than 1 week before surgery;
8. Any other circumstances that are considered unsuitable for study participation by attending physicians or investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-22 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting (PONV) within 24 hours following surgery | Up to 24 hours after surgery
  Nausea is diagnosed when the patient has gastrointestinal symptoms but does not vomit stomach contents. The severity of nausea is assessed using a digital subjective score scale (the scale ranges from 0 to 10, where 0 points represent no nausea, and 10 points represent the most severe nausea). Vomiting is diagnosed when the patient has gastrointestinal symptoms and retching or vomits gastric contents. Retching refers to the act of vomiting, but no stomach contents are vomited out.

SECONDARY OUTCOMES:
Incidence of PONV within 48 hours after surgery | Up to 48 hours after surgery
  Nausea is diagnosed when the patient has gastrointestinal symptoms but does not vomit stomach contents. The severity of nausea is assessed using a digital subjective score scale (the scale ranges from 0 to 10, where 0 points represent no nausea, and 10 points represent the most severe nausea). Vomiting is diagnosed when the patient has gastrointestinal symptoms and retching or vomits gastric contents. Retching refers to the act of vomiting, but no stomach contents are vomited out.
Incidence of complications within 30 days after surgery | Up to 30 days after surgery
  Postoperative complications are defined as new-onset medical events that are harmful to patients' recovery and required therapeutic intervention, i.e., grade II or above on the Clavien-Dindo classification.
Subjective sleep quality score within 3 days after surgery | Up to 3 days after surgery
  Subjective sleep quality was evaluated with the NRS (an 11-point scale where 0=the worst night sleep and 10=the best night sleep).
Incidence of emergence delirium (ED) | Up to 30 minutes after surgery or during the stay in PACU
  Delirium is assessed with the Confusion Assessment Method for the Intensive Care Unit. The assessments are performed at 10 minutes and 30 minutes after admission to the post-anesthesia care unit (PACU), or before leaving the PACU.
Incidence of delirium within 3 days after surgery | Up to 3 days after surgery
  Delirium is assessed with the Three-dimensional Confusion Assessment Method (3D-CAM) twice daily (between 8-10 am and 18-20 pm) during the first 3 days after surgery.
Length of stay in hospital after surgery | Up to 30 days after surgery
  Length of stay in hospital after surgery

OTHER OUTCOMES:
Incidence of intraoperative awareness | Up to 24 hours after surgery
  Intraoperative awareness is assessed with the modified Brice questionnaire during PACU stay and on the first postoperative day
Incidence of dreaming during general anesthesia | Up to 24 hours after surgery
  Assessed with the modified Brice questionnaire on the first day after surgery. Record whether the patient can recall the content of the dream (divided into clear, unclear, and forget) and the impact of the dream on the patient's subjective feelings (divided into pleasure, normal, sad, and nightmares)

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (10):
- China (10):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Hospital of the Ministry of Health, Beijing, Beijing Municipality
  - Beijing YouAn Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fuwai Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - Wuhan Puai Hospital, Wuhan, Hubei
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geng ZY, Liu YF, Wang SS, Wang DX. Intra-operative dexmedetomidine reduces early postoperative nausea but not vomiting in adult patients after gynaecological laparoscopic surgery: A randomised controlled trial. Eur J Anaesthesiol. 2016 Oct;33(10):761-6. doi: 10.1097/EJA.0000000000000491. PMID 27307217
- [Background] Dewinter G, Staelens W, Veef E, Teunkens A, Van de Velde M, Rex S. Simplified algorithm for the prevention of postoperative nausea and vomiting: a before-and-after study. Br J Anaesth. 2018 Jan;120(1):156-163. doi: 10.1016/j.bja.2017.08.003. Epub 2017 Nov 23. PMID 29397124
- [Background] Gan TJ, Diemunsch P, Habib AS, Kovac A, Kranke P, Meyer TA, Watcha M, Chung F, Angus S, Apfel CC, Bergese SD, Candiotti KA, Chan MT, Davis PJ, Hooper VD, Lagoo-Deenadayalan S, Myles P, Nezat G, Philip BK, Tramer MR; Society for Ambulatory Anesthesia. Consensus guidelines for the management of postoperative nausea and vomiting. Anesth Analg. 2014 Jan;118(1):85-113. doi: 10.1213/ANE.0000000000000002. PMID 24356162
- [Background] Li CJ, Wang BJ, Mu DL, Hu J, Guo C, Li XY, Ma D, Wang DX. Randomized clinical trial of intraoperative dexmedetomidine to prevent delirium in the elderly undergoing major non-cardiac surgery. Br J Surg. 2020 Jan;107(2):e123-e132. doi: 10.1002/bjs.11354. PMID 31903588
- [Background] Joo J, Park S, Park HJ, Shin SY. Ramosetron versus ondansetron for postoperative nausea and vomiting in strabismus surgery patients. BMC Anesthesiol. 2016 Jul 22;16(1):41. doi: 10.1186/s12871-016-0210-5. PMID 27449404
- [Background] Pym A, Ben-Menachem E. The effect of a multifaceted postoperative nausea and vomiting reduction strategy on prophylaxis administration amongst higher-risk adult surgical patients. Anaesth Intensive Care. 2018 Mar;46(2):185-189. doi: 10.1177/0310057X1804600207. PMID 29519221
- [Background] Burkhardt T, Czorlich P, Mende KC, Treitz A, Kiefmann R, Westphal M, Schmidt NO. Postoperative Nausea and Vomiting Following Craniotomy: Risk Factors and Complications in Context of Perioperative High-dose Dexamethasone Application. J Neurol Surg A Cent Eur Neurosurg. 2019 Sep;80(5):381-386. doi: 10.1055/s-0039-1685194. Epub 2019 May 10. PMID 31075810
- [Background] Laufenberg-Feldmann R, Muller M, Ferner M, Engelhard K, Kappis B. Is 'anxiety sensitivity' predictive of postoperative nausea and vomiting?: A prospective observational study. Eur J Anaesthesiol. 2019 May;36(5):369-374. doi: 10.1097/EJA.0000000000000979. PMID 30865002
- [Background] de Boer HD, Detriche O, Forget P. Opioid-related side effects: Postoperative ileus, urinary retention, nausea and vomiting, and shivering. A review of the literature. Best Pract Res Clin Anaesthesiol. 2017 Dec;31(4):499-504. doi: 10.1016/j.bpa.2017.07.002. Epub 2017 Jul 8. PMID 29739538
- [Background] Horn CC, Wallisch WJ, Homanics GE, Williams JP. Pathophysiological and neurochemical mechanisms of postoperative nausea and vomiting. Eur J Pharmacol. 2014 Jan 5;722:55-66. doi: 10.1016/j.ejphar.2013.10.037. Epub 2013 Oct 26. PMID 24495419
- [Background] Gan TJ, Belani KG, Bergese S, Chung F, Diemunsch P, Habib AS, Jin Z, Kovac AL, Meyer TA, Urman RD, Apfel CC, Ayad S, Beagley L, Candiotti K, Englesakis M, Hedrick TL, Kranke P, Lee S, Lipman D, Minkowitz HS, Morton J, Philip BK. Fourth Consensus Guidelines for the Management of Postoperative Nausea and Vomiting. Anesth Analg. 2020 Aug;131(2):411-448. doi: 10.1213/ANE.0000000000004833. PMID 32467512
- [Background] Grant MC, Kim J, Page AJ, Hobson D, Wick E, Wu CL. The Effect of Intravenous Midazolam on Postoperative Nausea and Vomiting: A Meta-Analysis. Anesth Analg. 2016 Mar;122(3):656-663. doi: 10.1213/ANE.0000000000000941. PMID 26332858
- [Background] Ahn EJ, Kang H, Choi GJ, Baek CW, Jung YH, Woo YC. The Effectiveness of Midazolam for Preventing Postoperative Nausea and Vomiting: A Systematic Review and Meta-Analysis. Anesth Analg. 2016 Mar;122(3):664-676. doi: 10.1213/ANE.0000000000001062. PMID 26516802
- [Background] Barends CRM, Absalom AR, Struys MMRF. Drug selection for ambulatory procedural sedation. Curr Opin Anaesthesiol. 2018 Dec;31(6):673-678. doi: 10.1097/ACO.0000000000000652. PMID 30124543
- [Background] Horiguchi Y, Ohta N, Yamamoto S, Koide M, Fujino Y. Midazolam suppresses the lipopolysaccharide-stimulated immune responses of human macrophages via translocator protein signaling. Int Immunopharmacol. 2019 Jan;66:373-382. doi: 10.1016/j.intimp.2018.11.050. Epub 2018 Dec 5. PMID 30530051
- [Background] Wesolowski AM, Zaccagnino MP, Malapero RJ, Kaye AD, Urman RD. Remimazolam: Pharmacologic Considerations and Clinical Role in Anesthesiology. Pharmacotherapy. 2016 Sep;36(9):1021-7. doi: 10.1002/phar.1806. Epub 2016 Sep 1. PMID 27496519
- [Background] Brice DD, Hetherington RR, Utting JE. A simple study of awareness and dreaming during anaesthesia. Br J Anaesth. 1970 Jun;42(6):535-42. doi: 10.1093/bja/42.6.535. No abstract available. PMID 5423844
- [Background] Hines S, Steels E, Chang A, Gibbons K. Aromatherapy for treatment of postoperative nausea and vomiting. Cochrane Database Syst Rev. 2018 Mar 10;3(3):CD007598. doi: 10.1002/14651858.CD007598.pub3. PMID 29523018